CLINICAL TRIAL: NCT06907914
Title: The Effect of Schroth Exercises on Scapular Muscle Activation in Children With Thoracic Hyperkyphosis
Brief Title: Schroth and Scapular Muscle Activation in Hyperkyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aza_isu2
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-04

CONDITIONS: Hyperkyphosis, Adolescent; Muscle Activation; Scapula; Deformity, Acquired; Exercise Therapy
Keywords: Spine; Schroth; sEMG; Physiotehrapy; Scapula; Thoracic Hyperkyphosis
MeSH Terms: conditions — Scheuermann Disease; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: the intervention group receiving Schroth exercises combined with postural education, and the control group receiving only postural education while placed on a waiting list. Both groups will be evaluated at baseline and after the 8-week intervention period
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will employ assessor and statistician blinding. The physiotherapists performing baseline and post-intervention assessments will be blinded to group allocation to minimize bias. Additionally, statistical analyses will be conducted by a researcher blinded to group assignments. Participants and therapists delivering the intervention will not be blinded due to the nature of the exercise-based intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in the experimental group will undergo a supervised 3D Schroth-based exercise program with postural education. The intervention will be applied 3 times per week for 8 weeks, totaling 24 sessions, each lasting approximately 45 minutes, delivered in-person by a trained physiotherapist.
  Exercises will include corrective postural training, scapular stabilization, rotational breathing, and static stretching. The program is delivered in two progressive phases:
  Weeks 1-4: Postural awareness and basic muscle activation
  Weeks 5-8: Functional integration and advanced stabilization
  Progression criteria are based on repetitions: exercises begin at 9 reps × 3 sets, and progress to 15 reps × 3 sets. Static stretches start with 20 seconds × 2 sets and are increased to 3 sets before progressing. All exercises are individualized based on clinical assessment.
  Interventions: Other: Schroth
- Group B (No Intervention): The control group will receive a single, standardized session of postural education at the beginning of the study, during which general information about correct posture, ergonomic principles, and spinal health will be provided. Following this session, participants in the control group will be placed on a waiting list and monitored for a period of 8 weeks. During this time, they will not receive any specific exercise intervention or additional therapeutic program related to posture or muscle strengthening. Regular follow-up will be conducted to ensure participant safety and to monitor any changes or adverse events throughout the waiting period.

INTERVENTIONS:
Other: Schroth — The Schroth intervention consists of a structured, three-dimensional exercise program based on scoliosis-specific principles. It incorporates corrective postural alignment, rotational breathing techniques, and targeted activation of spinal and scapular stabilizing muscles. The exercises are designed to improve postural control, enhance muscle endurance, and promote neuromuscular re-education for better functional alignment during daily activities.
  Arms: Group A

SUMMARY:
This randomized controlled trial aims to investigate the effects of Schroth exercises on scapular muscle activation in children with thoracic hyperkyphosis. A total of 56 participants will be randomly assigned to either the Schroth exercise group or the control group receiving postural education. The intervention group will complete an 8-week supervised Schroth program focusing on three-dimensional correction, rotational breathing, and postural awareness. Primary outcome is scapular muscle activation measured by surface EMG. Secondary outcomes include muscle strength, scapular endurance, kyphotic appearance, posture, and pain. The results will guide clinical management and preventive strategies for children with postural thoracic hyperkyphosis.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial aims to investigate the effects of Schroth-based three-dimensional exercises on scapular muscle activation in children with postural thoracic hyperkyphosis. Thoracic hyperkyphosis, commonly observed during childhood and adolescence, not only leads to spinal deformity but also negatively impacts scapular positioning, upper extremity function, and overall posture. Weakness and poor activation of scapular stabilizing muscles may contribute to the progression of kyphosis and functional limitations.

The Schroth method is a scoliosis-specific exercise approach designed to improve spinal alignment through three-dimensional postural correction, rotational breathing, and muscle stabilization techniques. Although widely used for spinal deformities such as scoliosis and kyphosis, its specific effects on scapular muscle activation remain insufficiently studied. This study will explore the potential of Schroth exercises to enhance scapular muscle function, which may contribute to improved posture, increased muscle strength and endurance, better scapular performance, reduced kyphotic appearance, and alleviation of pain.

The intervention group will participate in an 8-week supervised exercise program consisting of individualized Schroth exercises, focusing on postural awareness and scapular control during functional activities. By targeting scapular muscle activation, the study seeks to determine whether integrating Schroth exercises into physiotherapy practice can improve clinical outcomes and inform evidence-based approaches for managing postural thoracic hyperkyphosis in the pediatric population. Findings from this study may also contribute to developing preventive health strategies to protect musculoskeletal health in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic kyphosis angle (Cobb) between ≥40° and <70° on lateral radiographs
* Aged 7-18 years
* Risser stage 0-5, indicating ongoing skeletal development

Exclusion Criteria:

* Congenital or rigid spinal deformities/anomalies
* Major musculoskeletal surgery or trauma, especially involving the spine
* Physiotherapeutic intervention for the spine in the last 6 months
* Current brace use
* BMI ≥ 30
* Regular upper extremity sports involvement (e.g., swimming, volleyball) at least twice a week for one year
* More than 60 minutes of moderate-to-high intensity physical activity per week
* Visual impairments or light sensitivity
* Positive vestibular (Unterberger) test
* Hearing impairments
* Cognitive difficulties affecting comprehension
* Systemic diseases (diabetes, hypothyroidism, infection, malignancy)
* Neurological disorders
* Active rheumatic diseases

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Activation (sEMG) | 8 weeks
  Surface electromyography (sEMG) will assess the activation of the upper, middle, lower trapezius, and serratus anterior muscles, following SENIAM protocols. Signals will be normalized to %MVC and analyzed for concentric, isometric, and eccentric phases using RMS methods with a 20 Hz high-pass filter.

SECONDARY OUTCOMES:
Muscle Strength | 8 weeks
  Scapular stabilizing muscle strength will be measured using a handheld dynamometer (Lafayette Instrument). Higher force values (in Newtons) indicate greater muscle strength and improved functional capacity of the scapular muscles. An increase in the score reflects muscle strength gains, while a decrease indicates weakness or functional decline.
Scapular Muscle Endurance Test | 8 weeks
  Scapular muscle endurance will be evaluated using the Scapular Muscle Endurance Test, which measures the duration (in seconds) that scapular muscles can sustain an isometric contraction. A higher score indicates better endurance capacity, while a lower score reflects fatigue or reduced muscle endurance.
Kyphosis-Specific Spinal Appearance Questionnaire | 8 weeks
  The Kyphosis-Specific Spinal Appearance Questionnaire is a 10-item, 5-point Likert scale (range: 1 to 5 per item, total score range: 10 to 50) designed to assess patients' perception of their spinal appearance related to thoracic hyperkyphosis. Higher scores indicate worse perceived deformity and greater concern about appearance.
PostureScreen Mobile Application | 8 weeks
  Provides objective measurements of postural deviations. Improvements are indicated by reductions in deviation angles or distances.
Postural Habits and Awareness Scale | 8 weeks
  The Postural Habits and Awareness Scale consists of 19 items, each scored on a 5-point Likert scale (total score range: 19 to 95). Higher scores indicate better postural habits and awareness.
Numeric Rating Scale (NRS) | 8 weeks
  Pain intensity will be measured using the Numeric Rating Scale (NRS) during rest, physical activity, and at night. The scale ranges from 0 (no pain) to 10 (worst possible pain). A decrease in NRS scores indicates pain relief, while an increase signifies worsening pain.
Global Rating of Change (GROC) scale | 8 weeks
  Participant satisfaction with the intervention will be assessed using the Global Rating of Change (GROC) scale. The GROC is an 7-point scale ranging from -3 (very much worse) to +3 (completely recovered), with 0 indicating no change. Positive scores indicate perceived improvement, zero represents no change, and negative scores indicate worsening of symptoms or dissatisfaction with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Assoc Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Istanbul, Turkey (Türkiye)